CLINICAL TRIAL: NCT03130894
Title: Association Between Microbiota-dependent Metabolite Trimethylamine-N-oxide and Type 2 Diabetes
Brief Title: Association Between TMAO and Diabetes
Status: Completed | Type: Observational
Sponsor: Liegang Liu (Other)
Responsible Party: Sponsor-Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: 2012BAI02B02
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Type2 Diabetes
Keywords: trimethylamine-N-oxide; type2 Diabetes; enzyme flavin monooxygenase 3 polymorphisms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control: A FPG concentration < 6.1 mmol/l, and a 2-h oral glucose tolerance test (OGTT) plasma glucose concentration < 7.8 mmol/l was considered normal glucose tolerance.
  Interventions: Other: Plasma TMAO concentration
- Type 2 diabetes: Type 2 diabetes was diagnosed when fasting plasma glucose (FPG) ≥ 7.0 mmol/l, and/or 2-h post-glucose load ≥ 11.1 mmol/l.
  Interventions: Other: Plasma TMAO concentration

INTERVENTIONS:
Other: Plasma TMAO concentration — Plasma TMAO concentration

SUMMARY:
Background: The association of trimethylamine-N-oxide (TMAO), a microbiota dependent metabolite from dietary choline and carnitine, with type 2 diabetes was inconsistent.

Objective: The investigators planned to investigate the association between plasma TMAO and newly diagnosed type 2 diabetes as well as whether the association could be modified by the TMAO-generating enzyme flavin monooxygenase 3 (FMO3) polymorphisms.

Design: This is an age- and sex-matched case-control study of 2694 participants: 1346 newly diagnosed cases of type 2 diabetes and 1348 controls. The patients of newly diagnosed type 2 diabetes were consecutively recruited from those attending for the first time the outpatient clinics of Department of Endocrinology, Tongji Medical College Hospital, Wuhan, China, from 2012 January to December 2014. Concomitantly, the investigators recruited healthy individuals who were frequency-matched by age (±5 years) and sex to patients from an unselected population undergoing a routine health check-up in the same hospital. The inclusion criteria for controls and newly diagnosed type 2 diabetes were: age ≥ 30 years, body mass index (BMI) < 40 kg/m2, no history of a diagnosis of diabetes and no history of receiving pharmacological treatment for hyperlipidaemia or hypertension. Patients with clinically significant neurological, endocrinological or other systemic diseases, as well as acute illness or chronic inflammatory or infective diseases, were excluded from the study. All the participants enrolled were of Chinese Han ethnicity. All the participants gave informed written consent to the study and did not take any medication known to affect glucose tolerance or insulin secretion before participation. The study was approved by the ethics committee of the Tongji Medical College. Concentrations of plasma TMAO were measured, and FMO3 E158K polymorphism (rs2266782) were genotyped.

ELIGIBILITY:
Inclusion Criteria:

* Concomitantly, we recruited healthy individuals who were frequency-matched by age (±5 years) and sex to patients from an unselected population undergoing a routine health check-up in the same hospital.
* The inclusion criteria for controls and newly diagnosed type 2 diabetes were: age ≥ 30 years, body mass index (BMI) < 40 kg/m2, no history of a diagnosis of diabetes and no history of receiving pharmacological treatment for hyperlipidaemia or hypertension.

Exclusion Criteria:

* Patients with clinically significant neurological, endocrinological or other systemic diseases, as well as acute illness or chronic inflammatory or infective diseases, were excluded from the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the participants enrolled were of Chinese Han ethnicity. They gave informed written consent to the study and did not take any medication known to affect glucose tolerance or insulin secretion before participation.
Sampling Method: Probability Sample
Enrollment: 2694 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
type 2 diabetes | through recruitment completion, an average of 3 years
  odd ratio (OR) for type 2 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Liegang Liu, PhD, Study Director — Huazhong University of Science and Technology

REFERENCES:
- [Derived] Shan Z, Sun T, Huang H, Chen S, Chen L, Luo C, Yang W, Yang X, Yao P, Cheng J, Hu FB, Liu L. Association between microbiota-dependent metabolite trimethylamine-N-oxide and type 2 diabetes. Am J Clin Nutr. 2017 Sep;106(3):888-894. doi: 10.3945/ajcn.117.157107. Epub 2017 Jul 19. PMID 28724646